CLINICAL TRIAL: NCT03504462
Title: Specific Block of the Plantar Branches of the Tibial Nerve Under Ultrasound for Foot Surgery : A Monocentric Pilot Study
Brief Title: Feasibility of Specific Anesthesia of the Forefoot Preserving the Sensitivity of the Heel for Foot Surgery
Acronym: DISTIB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CMC Ambroise Paré (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2018/03
Record Dates: First submitted 2018-04-04; First posted 2018-04-20 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2019-12

CONDITIONS: Hallux Valgus and Bunion (Disorder); Morton Neuroma; Metatarsal Fracture; Ingrown Nail; Foot Wound; Foot Infection
Keywords: Foot surgery; Regional Anesthesia; Regional Analgesia; Ultrasound; Distal block; Plantar nerve block
MeSH Terms: conditions — Hallux Valgus; Bunion; Morton Neuroma; Nails, Ingrown; Foot Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Distal tibial nerve block (Experimental): Patient receiving a specific block of medial and lateral plantar nerves in order to preserve the calcaneal nerve
  Interventions: Procedure: Specific block of medial and lateral plantar nerves

INTERVENTIONS:
Procedure: Specific block of medial and lateral plantar nerves — Specific injection of long duration local anesthetic in contact with medial and lateral plantar nerves.
  Local anesthetic : Ropivacaine : 0,375% - 5 ml per nerve.

SUMMARY:
Foot surgery is a painful surgery that is usually scheduled in outpatients. A good management of analgesia is the crucial point. Regional anesthesia (RA) is the gold standard, that provides good anesthesia and a long duration of analgesia. The sciatic nerve block (or its branches) is the most adapted analgesic technique.

Limitation of proximal sciatic block is the motor block of the ankle and results in the impossibility, for the patient, to walk during the early post-operative period. Distal block of the sciatic nerve (tibial and fibular nerve blocks), at the level of the ankle, has been proposed to maintain the mobility of the ankle, to make deambulation with crutches easier. Nevertheless, the lack of sensibility of the heel remains a limitation for early walking, even with adapted shoes (ie : Barouk).

A specific anesthesia of the distal part of the foot, respecting the heel, could be the best option to provide an early deambulation and a suitable analgesia.

Ultrasound identification and specific anesthesia of the branches supplying the distal part of the foot (medial and lateral plantar nerves) could meet this dual objective : good anesthesia and suitable analgesia for early deambulation.

This study is a feasibility study of a specific block of the plantar branches of the tibial nerve, to preserve the sensibility of the heel, in case of foot surgery. The safety of the procedure will be assessed according to the rate of postoperative dysesthesia.

DETAILED DESCRIPTION:
Block of the medial and lateral plantar branches of the tibial nerve will be performed under the medial malleolar-calcaneal axis (MMCA) in order to preserve the calcaneal nerves.

Blocks of the deep peroneal nerve (DPN) and the superficial peroneal nerve (SPN) will be added to provide an adequate anesthesia.

Every block will be performed under Ultrasound using a 27-gauge, 5-cm, short bevel needle.

5 mL of 0.375% Ropivacaine will be injected for each block. The sensory blocks will be assessed by pinprick test and cold test every 10 minutes for 40 minutes in the following locations: Calcaneal nerves, Lateral plantar nerve and Medial plantar nerve.

The extent of sensory block will be graded as follows: 2: normal sensation; 1: decreased sensation; and 0: no sensation (complete block).

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a foot surgery
* Consent for participation
* Affiliation to the french social security system

Exclusion Criteria:

* Patient's refusal
* Existence of major spontaneous or acquired haemostatic disorders
* Infection at the point of puncture
* Allergy to local anesthetic or analgesic
* Pregnant or likely to be pregnant
* Patients under protection of the adults (guardianship, curator or safeguard of justice)
* Patients whose cognitive state does not allow assessment by the scales used
* Neuropathic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-06-25 (Actual); Primary Completion 2019-09-25 (Actual); Study Completion 2019-10-23 (Actual)

PRIMARY OUTCOMES:
Feasibility of a specific block of the lateral and medial plantar nerves | 40 minutes
  Pinprick and cold test on the sole of the foot - Cartography of the sole - Ipsilateral versus Contralateral test Numeric Scale for Pin-Prick test and Cold test : 2: normal sensation, 1: decreased sensation, 0: total loss of sensation

SECONDARY OUTCOMES:
Feasibility of the foot surgery with a specific block of the lateral and medial plantar nerves | 40 minutes
  Usage (or not) of an additional anesthetic procedure to perform the surgery
Ability to recognize plantar nerves under ultrasound | 40 minutes
  Numeric Rating Scale for Visualization : from 0 (very difficult) to 100 (very easy)
Patient satisfaction | At the end of surgery (2 hours maximum)
  Numeric Rating Scale for Satisfaction : from 0 (very unsatisfied) to 100 (very satisfied)
Patient comfort during block performance | 40 minutes
  Numeric Rating Scale for Pain : from 0 (no pain) to 100 (severe pain)
Complication | Day 15 and Day 30 After Surgery
  Questionnaire about toe mobility, foot sensitivity and potential sensory anomalies such as numbness, itching or tingling.

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien Bloc, MD, Principal Investigator — CMC Ambroise Paré
Locations (1):
- CMC Ambroise Paré, Neuilly-sur-Seine, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No